CLINICAL TRIAL: NCT02824354
Title: Multicentre, Randomised, Double-blind, Placebo-controlled Trial of Nalmefene in Patients With Alcoholic Compensated Cirrhosis for the Treatment of Alcohol Dependence.
Brief Title: Nalmefene in Patients With Alcoholic Compensated Cirrhosis for the Treatment of Alcohol Dependence.
Acronym: NalmeCir
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI2015_843_0017
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cirrhosis; Alcohol Dependence; Nalmefene
MeSH Terms: conditions — Fibrosis; Alcoholism | interventions — nalmefene; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): The placebo will have the same composition as the active treatment (without the drug substance) and an identical appearance. White, oval, biconvex, 6.0 x 8.75 mm film-coated tablet engraved with "S" on one side.
  Interventions: Drug: placebo
- Nalmefene (Experimental): Drug : 'Nalmefene (Selincro®) 18 mg tablet is a white, oval, biconvex, 6.0 x 8.75 mm film-coated tablet engraved with "S" on one side. It contains 18.06 mg nalmefene (in the form of hydrochloride dihydrate).
  Nalmefene must be taken as-needed: on each day the patient perceives a risk of drinking alcohol, one tablet should be taken, preferably 1-2 hours prior to the anticipated time of drinking. If the patient has started drinking alcohol without taking nalmefene, the patient should take one tablet as soon as possible.
  The maximum dose of nalmefene is one tablet per day. Nalmefene can be taken with or without food.
  Interventions: Drug: Nalmefene (Selincro®) 18 mg tablet

INTERVENTIONS:
Drug: Nalmefene (Selincro®) 18 mg tablet — Evaluate the efficacy, tolerability and safety of nalmefene for reduction of alcohol consumption (reduction of the number of monthly heavy drinking days, and daily total alcohol consumption) in alcohol-dependent patients with alcoholic compensated cirrhosis.
  Arms: Nalmefene
Drug: placebo — Evaluate the efficacy, tolerability and safety of nalmefene for reduction of alcohol consumption (reduction of the number of monthly heavy drinking days, and daily total alcohol consumption) in alcohol-dependent patients with alcoholic compensated cirrhosis.
  Arms: placebo

SUMMARY:
Nalmefene is the first drug to obtain Marketing Authorisation in France for reduction of alcohol consumption.

DETAILED DESCRIPTION:
Nalmefene is the first drug to obtain Marketing Authorisation in France for reduction of alcohol consumption. It appears to be significantly more effective in the group of heavy drinkers, while the mean alcohol consumption in studies conducted in cirrhotic patients is greater than 120 g/day.

No data are available concerning nalmefene in alcohol-dependent patients with alcoholic cirrhosis. However, nalmefene could represent an attractive alternative to reduce heavy drinking in patients with alcoholic cirrhosis, with potential improvement of liver function. No comparator is available for nalmefene, as all other molecules require abstinence prior to starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* the patient has signed and dated the informed consent form,
* blood alcohol concentration < 0.02% at the screening visit,
* alcohol-dependent patient according to DSM-IV-TR criteria ,
* patient with compensated cirrhosis (cirrhosis demonstrated by clinical and laboratory and/or morphological examinations and/or by a noninvasive test and/or by liver biopsy), Child A or B,
* patient with at least a high drinking risk level (a moderate risk level is defined as a consumption ≥ 60 g of alcohol/day for men and ≥ 40 g of alcohol/day for women),
* male or female, over the age of 18 years, excluding protected majors,
* patient with a stable address and telephone number,
* name and address of a family member who will be contacted in the event of loss of contact with the patient,
* women of childbearing potential:

  * must accept not to become pregnant during the study and,
  * must use an effective method of contraception (adequate contraception is defined as oral, systemic contraception, intrauterine device, diaphragm in combination with spermicide, or condom for the male partner in combination with spermicide) or,
  * must have had their last natural menstruation ≥ 24 months before the screening visit or,
  * must have been surgically sterilized before the screening visit or,
  * must have undergone hysterectomy before the screening visit or,
  * must have no sexual activity with a male partner
* patient covered by French national health insurance.

Exclusion Criteria:

* cirrhosis Child Pugh C (decompensated cirrhosis)
* cirrhosis complicated by hepatocellular carcinoma or type I or II hepatorenal syndrome or poorly controlled portal hypertension,
* severe acute alcoholic hepatitis, not responding to corticosteroids by the 7th day defined by a Lille model > 0.56 (www.lillemodel.com/score.asp)
* hepatic encephalopathy during the 6 months preceding the screening visit,
* patient with fewer than 6 heavy drinking days during the 4 weeks preceding the screening visit (a heavy drinking day is defined as alcohol consumption of ≥ 60 g/day for men, and ≥ 40 g/day for women),
* patient with at least 14 consecutive days of abstinence during the 4 weeks preceding the screening visit,
* patient with a CIWA-Ar score (Revised Clinical Institute Withdrawal Assessment for Alcohol) ≥ 10,
* patient with:
* a disorder other than alcohol or nicotine dependence, as evaluated on the MINI (Mini-International Neuropsychiatric Interview)
* antisocial personality disorder evaluated with the MINI questionnaire,
* other disorders for which treatment must take priority to the treatment of alcohol dependence, or which are likely to interfere with the study treatment or compromise adherence to treatment,
* cannabis use does not constitute an exclusion criterion except when it meets the criterion of cannabis dependence
* patient with a suicide risk evaluated using the suicidal tendency module of the MINI (the patient answers "Yes" to one of questions C2, C3, C4, C5 or C6 of the questionnaire),
* patient with a history of delirium tremens or alcohol withdrawal seizures,
* ongoing use of addictive substances other than cannabis, nicotine or benzodiazepines,
* presence of a disorder of comprehension, mental retardation or encephalopathy,
* presence of clinically significant unstable disease (e.g.: renal failure, cardiovascular, pulmonary, gastrointestinal, gastrointestinal, endocrine, neurological, infectious, neoplastic disease or metabolic disorders,
* clinically significant ECG abnormalities,
* history of serious drug allergy or hypersensitivity to nalmefene,
* ongoing or recent treatment (during the 3 months preceding the screening visit) with disulfiram, acamprosate, topiramate, naltrexone, carbimide, or opioid antagonists,
* ongoing or recent treatment (1 week preceding the screening visit) with opioid agonists or partial agonists,
* ongoing or recent treatment (8 weeks preceding the screening visit) with antipsychotics or antidepressants,
* patient taking or who has taken concomitant medications (see supplementary table),
* patient with another disease or taking medications, which, in the investigator's opinion, could interfere with evaluations of safety, tolerability and efficacy,
* treatment with an investigational medicinal product during the 30 days preceding the screening visit,
* ongoing or recent participation (during the 4 weeks preceding the screening visit) in a drinking disorders treatment or support programme, including Alcoholics Anonymous, disintoxication treatment and treatment of alcohol withdrawal symptoms,
* pregnancy or breastfeeding,
* patient who, in the investigator's opinion, has little chance of complying with the protocol or unsuitable for the study for any other reason,
* patient who has already participated in a clinical trial on nalmefene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Reduction of the number of monthly heavy drinking days after 6 months of treatment compared to baseline. | 6 months

SECONDARY OUTCOMES:
The number of non-drinking days during the treatment period; nalmefene arm versus placebo arm, | 6 months
Evaluation of craving; nalmefene arm responders versus nalmefene arm non-responders | 6 months
  Severity of Alcohol Dependence Questionnaire, Obsessive Compulsive Drinking Scale
Course of liver function after 6 months of treatment compared to baseline | 6 months
  • Course of liver function after 6 months of treatment compared to baseline:
  - nalmefene arm versus placebo arm, nalmefene arm responders versus nalmefene arm non-responders : - nalmefene arm versus placebo arm; - nalmefene arm responders versus nalmefene arm non-responders, PT, Bilirubin, ALT, GGT, Albumin, Creatinine. MELD and Child-Pugh scores
6 months survival | 6 months
  6-month survival: nalmefene arm versus placebo arm; nalmefene arm responders versus nalmefene arm non-responders

CONTACTS AND LOCATIONS:
Overall Officials: Eric NGUYEN-KHAC, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France